CLINICAL TRIAL: NCT03129893
Title: Ventilator Associated Complications in Neonate and Small Infant Undergoing Cardiac Surgery Using Cuffed and Uncuffed Tracheal Tubes. The PICU-BG-TT Study
Brief Title: Cuffed Versus Uncuffed Tracheal Tubes in PICU (PICU-BG-TT Study)
Acronym: PICU-BG-TT
Status: Completed | Type: Observational
Sponsor: FROM- Fondazione per la Ricerca Ospedale di Bergamo- ETS (Other)
Responsible Party: Sponsor
Other Study IDs: PICU-BG-TT
Record Dates: First submitted 2017-03-01; First posted 2017-04-26 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Intubation; Pediatric Surgery

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

GROUPS / COHORTS (2):
- Patients intubated with uncuffed tracheal tubes: Portex uncuffed TT sizes selected according to local institutional guidelines. Tracheal intubation performed under direct laryngoscopy by the oral or nasal route, without or with the use of bougies or stylets. TT insertion depth managed according to institutional guidelines in uncuffed TTs.
- Patients intubated with cuffed tracheal tubes: Cuffed TT sizes selected as follows: ID 3.0 mm for birth (>3 kg body weight) to < 8 months; ID 3.5 mm for 8 to < 12 months (Salgo, Schmitz et al. 2006). Tracheal intubation performed under direct laryngoscopy by the oral or nasal route, without or with the use of bougies or stylets. TT insertion depth managed according to the depth marking in cuffed TTs.
  Interventions: Device: Cuffed tracheal tubes

INTERVENTIONS:
Device: Cuffed tracheal tubes — Cuffed tracheal tube with an anatomically designed high volume - low pressure tube cuff, with a recommendation chart for tube size selection available for pediatric anesthesia
  Groups: Patients intubated with cuffed tracheal tubes

SUMMARY:
The CDC definition was used to identify patients with VAP and VAT. The CDC definition of VAP for infants < 1 y.o. and children > 1 or < 12 y.o. are based on clinical and X-ray criteria. The CDC definition of Tracheitis are based on absence of clinical and radiographic evidence of pneumonia and the following criteria: positive culture obtained by deep tracheal aspirate and 2 signs of symptoms with no recognizable cause [such as fever (>38.5°C), cough, new or increased sputum production, rhonchi, or wheezing].

The new CDC definition is used to identify patients with VAC and IVAC. The new definitions includes all associated complications (infection included) related to mechanical ventilation and exclude X-ray criteria.

VAP, VAT, VAC, IVAC rate, expressed as the number of VAP/VAT/VAC/IVAC episodes per 1000 mechanical ventilator days (VAP/1000 MV days), were calculated for phase 1 and phase 2.

DETAILED DESCRIPTION:
Ventilator associated pneumoniae (VAP) occurs in 9-27% of all intubated patients and is associated to an important morbidity and mortality. It is a serious complication among neonates and pediatric patients after cardiac surgery accounting for 6.8-32.2% of health-care associated infections. Ventilator associated tracheobronchitis (VAT) is common in adults and it has been described as a risk factor for the development of VAP. Studies have shown that treatment of VAT is associated with a lower rate of VAP and a lower mortality in adult patients. VAT has also been described in premature infants and children but it has been less studied than in adults.Recently, the Centers for Disease Control and Prevention (CDC) rolled out new surveillance definitions for patients receiving mechanical ventilation to be more objective and to render the data easier to collect and verify. The terms include ventilator-associated condition (VAC) and infection-related, ventilator-associated complication (IVAC). Studies in adults demonstrated that the VAC assessment was faster, more objective, and a superior predictor of outcomes. However, this approach has not yet been applied systematically to infants and children.For more than 50 years, uncuffed tracheal tubes have been commonly used for intubation in children under 8 years of age because of the anatomy of the pediatric larynx and the fear that the cuff will cause airway mucosal injury, leading to subglottic stenosis. However, since 2009, it is registered and available a new cuffed tracheal tube (TT) with an anatomically designed high volume-low pressure tube cuff, with a recommendation chart for tube size selection has recently become available for pediatric anesthesia.Weiss and colleagues enrolled 2246 patients in a randomized multi-centre trial and reported no increase of risk for post-extubation stridor with the use of the new microcuffed.Considering that microaspiration of contaminated oral secretions is one of the mechanisms leading to VAP and VAT, the use of cuffed TTs may be beneficial in VAP prevention as the superior tracheal seal may decrease the incidence of micro-aspiration. However, no study evaluated the incidence of VAP with the use of cuffed tracheal tubes is published since now.Despite of these new evidence, the use of uncuffed tube in neonatal and pediatric critical care still remain very common to minimize minor complications (i.e. mucosal damage due to the cuff), and consequently the use of cuffed or uncuffed tubes is equally recommended.The management of anesthesia according to standards procedures of the Bergamo anesthesia department is shifting from the uncuffed tubes only to microcuffed tubes, and it is aim of the present study to monitor this transition measuring the performance of the two TTs in terms of incidence of VAP and VAT (according to the CDC old definition) and in term of incidence of VAC and IVAC (according to CDC new definition).The CDC definition was used to identify patients with VAP and VAT. The CDC definition of VAP for infants < 1 y.o. and children > 1 or < 12 y.o. are based on clinical and X-ray criteria. The CDC definition of Tracheitis are based on absence of clinical and radiographic evidence of pneumonia and the following criteria: positive culture obtained by deep tracheal aspirate and 2 signs of symptoms with no recognizable cause [such as fever (>38.5°C), cough, new or increased sputum production, rhonchi, or wheezing].

The new CDC definition is used to identify patients with VAC and IVAC. The new definitions includes all associated complications (infection included) related to mechanical ventilation and exclude X-ray criteria.

VAP, VAT, VAC, IVAC rate, expressed as the number of VAP/VAT/VAC/IVAC episodes per 1000 mechanical ventilator days (VAP/1000 MV days), were calculated for phase 1 and phase 2.

ELIGIBILITY:
Inclusion Criteria:

* Neonates >35/40 gestation;
* Expected to require ventilation for > 24 hours;
* Age: 0 - 5 year.

Exclusion Criteria:

• Parents refused consent.

Max Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric patient in need intubation for cardiac surgery and transferred to the PICU.
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2017-01-01 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
The incidence rate difference of VAP and VAT between microcuffed TTs and uncuffed TTs | At PICU discharge, an average of 2 weeks
  The incidence rate difference of VAP and VAT between microcuffed TTs and uncuffed TTs

SECONDARY OUTCOMES:
The incidence rate difference of VAC and IVAC | At PICU discharge, an average of 2 weeks
  The incidence rate difference of VAC and IVAC
The reintubation rates for leakage | At PICU discharge, an average of 2 weeks
  The reintubation rates for leakage
The post-extubation airway morbidity (post-extubation stridor) | At PICU discharge, an average of 2 weeks
  The post-extubation airway morbidity (post-extubation stridor)
The duration of intubation | At PICU discharge, an average of 2 weeks
  The duration of intubation
The length of PICU stay | At PICU discharge, an average of 2 weeks
  The length of PICU stay

CONTACTS AND LOCATIONS:
Overall Officials: Mirco Nacoti, MD, Principal Investigator — ASST Papa Giovanni XXIII di Bergamo
Locations (1):
- Pediatric intensive care unit - ASST Papa Giovanni XXIII, Bergamo, BG, Italy

IPD SHARING:
Plan to Share IPD: No